CLINICAL TRIAL: NCT05898269
Title: Evaluation of the Diagnostic Performance of 4 Dynamic Tests Evaluating Preload Dependence in Patients With Acute Respiratory Distress Syndrome in the Prone Position
Brief Title: Fluid Responsiveness Prediction During Prone Position
Acronym: PROLOAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0315; 2023-A00920-45 (Other: ANSM)
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; Fluid responsiveness; Fluid resuscitation; Cardiac output; Cardiac preload; Prone position; Continuous cardiac output monitoring
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- Trendelenburg maneuver-EE OCC-EI OCC-Tidal volume challenge (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Trendelenburg maneuver-EE OCC-Tidal volume challenge-EI OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Trendelenburg maneuver-Tidal volume challenge-EI OCC-EE OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Trendelenburg maneuver-Tidal volume challenge-EE OCC-EI OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Trendelenburg maneuver-EI OCC-Tidal volume challenge-EE OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Trendelenburg maneuver-EI OCC-EE OCC-Tidal volume challenge (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EE OCC-EI OCC-Tidal volume challenge-Trendelenburg maneuver (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EE OCC-EI OCC-Trendelenburg maneuver-Tidal volume challenge (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EE OCC-Tidal volume challenge-Trendelenburg maneuver-EI OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EE OCC-Tidal volume challenge-EI OCC-Trendelenburg maneuver (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EE OCC-Trendelenburg maneuver-Tidal volume challenge-EI OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EE OCC-Trendelenburg maneuver-EI OCC-Tidal volume challenge (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EI OCC-Tidal volume challenge-EE OCC-Trendelenburg maneuver (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EI OCC-Tidal volume challenge-Trendelenburg maneuver-EE OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EI OCC-Trendelenburg maneuver-EE OCC-Tidal volume challenge (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EI OCC-Trendelenburg maneuver-Tidal volume challenge-EE OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EI OCC-EE OCC-Trendelenburg maneuver-Tidal volume challenge (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- EI OCC-EE OCC-Tidal volume challenge-Trendelenburg maneuver (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Tidal volume challenge-EI OCC-EE OCC-Trendelenburg maneuver (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Tidal volume challenge-EI OCC-Trendelenburg maneuver-EE OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Tidal volume challenge-Trendelenburg maneuver-EE OCC- EI OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Tidal volume challenge-Trendelenburg maneuver- EI OCC-EE OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Tidal volume challenge-EE OCC-Trendelenburg maneuver- EI OCC (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)
- Tidal volume challenge-EE OCC- EI OCC-Trendelenburg maneuver (Experimental): All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus.
  There are 24 different possibilities of sequence
  Interventions: Diagnostic Test: Trendelenburg maneuver; Diagnostic Test: End-expiratory occlusion test (EE OCC); Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC); Diagnostic Test: Tidal volume challenge; Diagnostic Test: Fluid bolus (reference diagnostic method)

INTERVENTIONS:
Diagnostic Test: Trendelenburg maneuver — Bed tilting from the +13° position to the -13° position for 60 seconds. Evaluator: relative change in continuous cardiac index between baseline, and the highest value observed during the maneuver
Diagnostic Test: End-expiratory occlusion test (EE OCC) — End-expiratory pause performed on the ventilator, and maintained for 15 seconds.
  Evaluator: relative change in continuous cardiac index between baseline, and the value observed in the last 5 seconds of the respiratory pause
Diagnostic Test: End-expiratory and end-inspiratory occlusion test (EI OCC) — End-inspiratory pause performed on the ventilator, and maintained for 15 seconds.
  Evaluator: relative change in continuous cardiac index between baseline, and the value observed in the last 5 seconds of the respiratory pause. The evaluator is calculated as the sum of the relative change in cardiac index observed during the end-expiratory pause and that of the end-inspiratory pause. Hence, for this test, the evaluator will be coupled with that of intervention 2 (end-expiratory occlusion test).
Diagnostic Test: Tidal volume challenge — Increase in tidal volume set on the ventilator from 6 ml.kg-1 of predicted body weight, to 8 ml.kg-1 for 60 seconds.
  Evaluator: difference in the pulse pressure variation measured at 6 ml.kg-1 and at 8 ml.kg-1.
Diagnostic Test: Fluid bolus (reference diagnostic method) — After the 4 tests, the patient will receive a 500-ml fluid bolus of crystalloids in less than 15 minutes.
  Evaluator (reference method): cardiac index measured by transpulmonary thermodilution before and immediately after the fluid bolus. Patients with a relative change in cardiac index > 15% will be identified as being fluid responders, and the others as non-responders.

SUMMARY:
Predicting fluid responsiveness is primordial when caring for patients with circulatory shock as it allows correction of preload-dependent low cardiac output states, while preserving patients of the deleterious effects of excessive fluid resuscitation.

Patients with severe acute respiratory distress syndrome (ARDS) treated with prone positioning (PP) are a specific subset of patients, as 1) they frequently present with shock; 2) excessive fluid administration may lead to respiratory worsening due to increased hydrostatic oedema with potential subsequent worse clinical outcome; and 3) all available dynamic tests evaluating fluid responsiveness can only be performed in patients in the supine condition (which in the case of severe ARDS patients in PP occurs only for 8h over 24h). These elements warrant the development of specific tests allowing the clinician to predict fluid responsiveness with enough exactitude when caring for these patients.

We hypothesize that there exists diagnostic heterogeneity in the predictive performance of 4 clinical tests to identify fluid responsiveness in ARDS patients in PP. For the matter of this study, these 4 tests are the Trendelenburg maneuver, the end-expiratory occlusion test, the end-expiratory occlusion test associated with the end-inspiratory occlusion test, and the tidal volume challenge. The diagnostic reference of the study will be the relative change in cardiac index measured by transpulmonary thermodilution before and after a 500 ml fluid bolus, and will allow the adjudication of patients as being fluid responsive or not.

The primary objective of the study is to determine the area under the ROC curve of each of the 4 tests, with their respective 95% confidence interval.

All enrolled patients will perform the 4 tests following a cross-over design and in a randomized sequence, separated by 1-min wash-out periods with return to hemodynamic baseline values, and concluded with the 500-ml fluid bolus. Patients will only participate once. The expected duration of study participation is 30 minutes maximum.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (including patient under protective measures/wardship)
* with ARDS as defined by the Berlin criteria
* in the prone position as per international guidelines
* with a calibrated continuous cardiac output monitoring device
* with a clinical indication for a fluid bolus as prescribed by the clinician in charge, and fulfilling at least 2 clinical criteria: mottles, tachycardia, hypotension, drop in cardiac output, oliguria, high arterial lactate concentration, or any other detailed criterion
* with no respiratory efforts

Exclusion Criteria:

* acute cor pulmonale
* patient treated with veno-venous extra-corporeal membrane oxygenation
* hemorrhagic shock
* Child-Pugh C cirrhosis
* death expected to occur in less than 24h
* decision to withhold or suspend active treatments
* intracranial hypertension
* lower limb amputation
* obstruction of the inferior vena cava
* acute abdominal syndrome
* absence of consent to participate
* pregnancy
* patient previously enrolled in the same study
* lack of affiliation to a social security regimen, as per French legislation
* patient deprived of its liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve (AUROC) of the evaluated tests. | 30 minutes
  The AUROC will be determined for each of the 4 clinical tests evaluated in this study. The reference method to define the AUROC to design the curve will be the fluid responsive status (responder vs. non-responder) as determined by the fluid bolus. For each test, the AUROC will be accompanied with its 95% confidence interval.

SECONDARY OUTCOMES:
Comparison of diagnostic performance of the evaluated tests. | 30 minutes
  For this outcome measure, the AUROCs will be determined as for the primary outcome measure. The AUROCs will be compared using the Delong's method, with adjustments for the repetition of measurements in a single patient.
Diagnostic performance metrics of each test | 30 minutes
  Sensitivity, specificity, positive predictive value, negative predictive value and likelihood ratios of the evaluated tests, computed for the optimal diagnostic threshold determined using the Youden J index of the ROC curve. The optimal threshold will only be computed for AUROCs significantly different from 0.5.
Weighted diagnostic performance of each test | 30 minutes
  Sensitivity, specificity, positive predictive value, negative predictive value and likelihood ratios of the evaluated tests, computed for the optimal diagnostic threshold determined using the Youden J index of the ROC curve, and adjusted using weighting based on the clinical tradeoff of the subsequent fluid bolus on hemodynamic benefit vs. the respiratory risk. The optimal threshold will only be computed for AUROCs significantly different from 0.5.
Grey zone area of the optimal diagnostic threshold of each test | 30 minutes
  Determination of the boundaries of a grey zone around the value of the optimal threshold of each test, in which the diagnostic performance is deemed clinically insufficient (excessive misclassification risk due to lack of discrimination). The grey zone around the optimal threshold will only be computed for AUROCs significantly different from 0.5.

CONTACTS AND LOCATIONS:
Overall Officials: Hodane YONIS, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Hôpital de la Croix Rousse, Hospices Civils de Lyon, Lyon
  - CHU de Nice - l'Archet 1, Nice
  - CHU Nice - Pasteur 2, Nice